CLINICAL TRIAL: NCT03690375
Title: A Prospective, Randomized, Split-Arm Pilot Study Investigating the Efficacy and Safety of Sciton's Broad Band Light for Improving the Clinical Signs of Senile Purpura
Brief Title: Broad Band Light for the Treatment and Prevention of Senile Purpura
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Siperstein Dermatology (Other)
Collaborators: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Purpura001
Record Dates: First submitted 2018-09-22; First posted 2018-10-01 (Actual); Results first posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2019-11

CONDITIONS: Senile Purpura; Bateman's Purpura
Keywords: skin atrophy; broad band bight; ecchymosis; collagen; elastin; RNA
MeSH Terms: conditions — Ecchymosis; Aortic Stenosis, Supravalvular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- BBL Left (Experimental): Left arm selected to be treated with BBL, right arm not treated
  Interventions: Device: Broad Band Light (BBL)
- BBL Right (Experimental): Right arm selected to be treated with BBL, left arm not treated
  Interventions: Device: Broad Band Light (BBL)

INTERVENTIONS:
Device: Broad Band Light (BBL) — Sciton's BBL treatment using a new protocol that utilizes a 590nm, 560nm, and skintyte filter

SUMMARY:
There will be five subjects over the age of 65, each with at least one ecchymotic lesion on each arm measuring at least one cm, and five control subjects under the age of 35, both who will be randomized to undergo 4 Sciton Broad Band Light (BBL) treatments on either their left or right arm one week apart. Subjects will fill out questionnaires, have pictures of their lower arms taken, and will be graded and measured by evaluators regarding the number and size of their ecchymoses as well as side effects such as blistering, pain, erythema, and swelling. One day after their 4th treatment on each arm, subjects will have biopsies done to be analyzed for changes in histology and gene expression. The subjects will follow up 1 month after their last treatments for final pictures of their lower arms and evaluations.

DETAILED DESCRIPTION:
This will be a single center, prospective, split-arm clinical study in which subjects will be randomized to which arm will be treated with Sciton's broad band light (BBL) treatment. All subjects will have their arms shaved prior to the procedure and cleaned thoroughly with alcohol. After the procedure a zinc-based sunscreen will be applied to both arms.

Before each of the four treatments, and 1 month after the last treatment, the subjects' number and square area of ecchymoses will be measured by an evaluator and photographs will be taken. Side effects will be measured the same day as the treatment as well as 1 day, 2 days, and 7 days after the first treatment.

A final assessment will be done by taking two skin biopsies from the subjects with senile purpura, one on treated skin and one on untreated skin, and one skin biopsy on untreated skin in the younger controls. The skin specimens will be bisected and one half will be submerged immediately in 10x volumes of formalin while the other half of the biopsy will be submerged immediately in 10x volumes of RNAlater (Thermo Fisher Scientific, Waltham, MA). These specimens will then be coded and sent to blinded evaluators that will embed half in paraffin sections and then stain them with hematoxylin and eosin (H&E), von Giesen and or periodic acid-Schiff (PAS).

Epidermal thickness will be measured on H&E-stained sections using the AxioVision image analysis software (Carl Zeiss Microimaging, Thornwood, NY). The epithelial thickness may vary from area to area within the biopsy. The thickness of the epithelium in µm will be measured at 6 points in each biopsy and averaged. Von Giesen-stained sections will be examined for elastosis, and PAS-stained sections will be examined for collagen.

Total RNA will be extracted using TRIzol Reagent (Thermo Fisher Scientific, Waltham, MA) and the RNeasy mini kit (Qiagen, Valencia, CA). RNA will be reverse transcribed using qScript™ cDNA Synthesis Kit (QuantaBio, Beverly, MA). Real-time qPCR reactions will be carried out using PerfeCTa SYBR® Green SuperMix (QuantaBio, Beverly, MA) in triplicates. Gene expression levels will be normalized to a housekeeping gene, and analyzed using t test of means and SEM. Potential analysis include various biomarkers for dermal remodeling (e.g., collagen type I, elastin), epidermal differentiation (e.g., keratin 1, filaggrin), and vascular changes (e.g., endothelin, Ang).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, aged >22
* In good general health as evidenced by medical history
* Ecchymosis greater than 1cm on each arm for the group with senile purpura

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Subjects with a history of any arm swelling
* Subjects with allergies to light
* Subjects with auto-immune skin conditions such as lupus, or vitiligo
* Subjects using topical retinol within the last 3 months
* Subjects with any scheduled laser, light, or surgical procedures on the arm during the study
* Subjects unwilling or unable to keep their arms still during digital pictures
* Subjects who are pregnant or nursing
* Subjects with a history of herpes simplex or zoster on their arms
* Subjects with current skin infections, tumors, or dermatitis on the arm
* Subjects with allergies to lidocaine
* Subjects with a history of keloid formation
* Subjects with a history of a bleeding disorder
* Subjects with allergies to adhesives

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Siperstein, MD, Study Director — Siperstein Dermatology/ University of Miami
Locations (1):
- Siperstein Dermatology Group, Boynton Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Faucz LL, Will SE, Rodrigues CJ, Hesse H, Moraes AC, Maria DA. Quantitative evaluation of collagen and elastic fibers after intense pulsed light treatment of mouse skin. Lasers Surg Med. 2018 Jan 16. doi: 10.1002/lsm.22782. Online ahead of print. PMID 29336034
- [Background] Bitter PH. Noninvasive rejuvenation of photodamaged skin using serial, full-face intense pulsed light treatments. Dermatol Surg. 2000 Sep;26(9):835-42; discussion 843. doi: 10.1046/j.1524-4725.2000.00085.x. PMID 10971556
- [Background] McKenzie NE, Saboda K, Duckett LD, Goldman R, Hu C, Curiel-Lewandrowski CN. Development of a photographic scale for consistency and guidance in dermatologic assessment of forearm sun damage. Arch Dermatol. 2011 Jan;147(1):31-6. doi: 10.1001/archdermatol.2010.392. PMID 21242389
- [Background] DeFatta RJ, Krishna S, Williams EF 3rd. Pulsed-dye laser for treating ecchymoses after facial cosmetic procedures. Arch Facial Plast Surg. 2009 Mar-Apr;11(2):99-103. doi: 10.1001/archfacial.2008.538. PMID 19289681
- [Background] Brauer JA, Farhadian JA, Bernstein LJ, Bae YS, Geronemus RG. Pulsed Dye Laser at Subpurpuric Settings for the Treatment of Pulsed Dye Laser-Induced Ecchymoses in Patients With Port-Wine Stains. Dermatol Surg. 2018 Feb;44(2):220-226. doi: 10.1097/DSS.0000000000001255. PMID 28858925
- [Background] Chang AL, Bitter PH Jr, Qu K, Lin M, Rapicavoli NA, Chang HY. Rejuvenation of gene expression pattern of aged human skin by broadband light treatment: a pilot study. J Invest Dermatol. 2013 Feb;133(2):394-402. doi: 10.1038/jid.2012.287. Epub 2012 Aug 30. PMID 22931923
- [Background] Prieto VG, Sadick NS, Lloreta J, Nicholson J, Shea CR. Effects of intense pulsed light on sun-damaged human skin, routine, and ultrastructural analysis. Lasers Surg Med. 2002;30(2):82-5. doi: 10.1002/lsm.10042. PMID 11870785

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 subjects with senile pupura were enrolled in the trial and analyzed. An additional 5 subjects without senile purpura were also enrolled as a control for some secondary measures.
Units Other Than Participants: arms
Groups:
- BBL Treatment: One arm was randomly selected to receive treatment with Sciton's BBL according to a protocol with multiple passes with different filters and settings.
- No Treatment: One arm was not treated
Period: Overall Study
Arm/Group | BBL Treatment | No Treatment
Started (While 10 subjects were enrolled, only 5 subjects were analyzed for senile purpura while the other 5 subjects were used as controls in some secondary measures) | 10; 10 arms | 10; 10 arms
Completed | 10; 10 arms | 10; 10 arms
Not Completed | 0; 0 arms | 0; 0 arms

BASELINE CHARACTERISTICS:
Population: The overall number of units analyzed represent the arms of participants with senile purpura.
Units Other Than Participants: arms
Groups:
- BBL Treatment: One arm was randomly selected to receive treatment with Sciton's BBL with multiple passes using a new protocol with varying filters and settings.
- Total: Total of all reporting groups
Arm/Group | BBL Treatment | No Treatment | Total
Number analyzed (Participants) | 10 | 10 | 10
Number analyzed (arms) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 5 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only the subjects with senile purpura (5 of 10) were analyzed for measurements of senile purpura
  Participants
    Female | 8 | 8 | 16
    Male | 2 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10
Square Area of Purpuric Lesions [Mean (Full Range); unit: cm2] — Measurement of purpuric lesion size was done by multiplying the width by the height of the lesion in cm and therefore the final measurement is cm2. This was done only in the 10 arms (5 participants) that had senile purpura at baseline. Population: Measurement of purpuric lesion size was only done in 10 arms (5 participants with senile purpura). The other 5 participants were used as controls for other measures.
  cm2
    number analyzed (Participants) | 5 | 5 | 5
    (all) | 22.8 [1 to 64.25] | 17.05 [1 to 51.25] | 19.925 [1 to 64.25]
Number of Purpuric Lesions [Mean (Full Range); unit: purpuric lesions] — The number of individual purpuric lesions were counted Population: Only 5 participants (10 arms) were analyzed regarding number of purpuric lesions and size of purpuric lesions. The additional 5 younger subjects were used as to compare changes in mrna and skin thickness but could not be used to measure purpuric lesions as they did not have any.
  purpuric lesions
    number analyzed (Participants) | 5 | 5 | 5
    (all) | 5.8 [1 to 9] | 5 [1 to 12] | 5.4 [1 to 12]

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline to 30 Days After the Last Treatment in the Number of Senile Purpura Lesions
Description: The number of purpuric lesions 30 days after the last treatment will be subtracted from the number of purpuric lesions at baseline
Time Frame: 51 days (Treatments done every 7 days starting on Day 0 and ending on Day 21, then the final outcome was measured 30 days after the last treatment)
Population: This outcome measure was only assessed in those with purpuric lesions
Measure: Median (Full Range); unit: number of purpuric lesions
Groups:
- BBL Treatment: One arm was randomly selected to receive treatment with Sciton's BBL
Arm/Group | BBL Treatment | No Treatment
Number analyzed (Participants) | 5 | 5
number of purpuric lesions | -3.55 [-12.75 to 0.75] | -.35 [-8.75 to 4]

2. Primary Outcome: The Change in Total Square Size of Purpuric Lesions From Baseline to 30 Days After the Last Treatment
Description: The size of the purpuric lesions will be measured by multiplying the height by the width in cm of each lesion and totaling the total cm2 area for each lesion on each arm. Then the total square area 30 days after the last treatment will be subtracted from the total square area at baseline.
Time Frame: 51 Days (30 days after the final treatment at Day 21)
Population: This measure was only assessed in those with purpuric lesions
Measure: Mean (Full Range); unit: cm2
Arm/Group | BBL Treatment | No Treatment
Number analyzed (Participants) | 5 | 5
cm2 | -4.8 [-12.75 to 0.75] | 9.95 [-4 to 55]

3. Secondary Outcome: Epidermal Thickness 1 Day After the Fourth BBL Treatment
Description: Measurement of epidermal thickness in um as measured by H&E stained sections using the AxionVision image analysis software based on slides from biopsies taken from the subjects 1 days after their last treatment.
Time Frame: 22 days (1 day after final treatment at day 21)
Population: Data collected for those participants with senile purpura for both interventions, data collected for those participants without for only the control no treatment arm
Measure: Mean (Full Range); unit: um
Groups:
- BBL Treatment Senile Purpura: One arm was randomly selected to receive treatment with Sciton's BBL in those with senile purpura
- No Treatment Senile Purpura: One arm was not treated in those with senile purpura
- No Treatment No Senile Purpura: Younger control participants without senile purpura
Arm/Group | BBL Treatment Senile Purpura | No Treatment Senile Purpura | No Treatment No Senile Purpura
Number analyzed (Participants) | 5 | 5 | 5
um | 54.89 [41.07 to 72.88] | 45.31 [25.29 to 70.40] | 53.82 [48.48 to 58.47]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | BBL Treatment | No Treatment
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

LIMITATIONS AND CAVEATS:
Small pilot study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/75/NCT03690375/Prot_SAP_001.pdf